CLINICAL TRIAL: NCT03788200
Title: Randomized, Controlled Trial of Posterior C1-2 Fusion Versus Bracing Alone for Treatment of Type II Odontoid Process Fractures in the Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018Kepler
Record Dates: First submitted 2018-12-26; First posted 2018-12-27 (Actual); Last update posted 2018-12-28 (Actual); Status verified 2018-12

CONDITIONS: Odontoid Fracture
MeSH Terms: interventions — Braces

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- post-injury bracing with rigid cervical collar (Active Comparator): Treatment arm #1 (8 weeks of post-injury bracing with rigid cervical collar): Participants randomized to this treatment arm will be treated with 8 weeks in a rigid cervical collar.
  Interventions: Procedure: Bracing
- posterior C1-2 instrumented fusion (Active Comparator): Participants randomized to this treatment arm will undergo posterior C1-2 instrumented fusion with either local bone grafting or autologous iliac crest bone grafting with or without allograft bone grafting. Bone grafting decision will be made by the treating surgeon. All remaining decisions surrounding medical and surgical care will be made by the attending spine surgeon involved in each case.
  Interventions: Procedure: posterior C1-C2 instrumented fusion

INTERVENTIONS:
Procedure: Bracing — Treatment arm #1 (8 weeks of post-injury bracing with rigid cervical collar): Participants randomized to this treatment arm will be treated with 8 weeks in a rigid cervical collar.
  Arms: post-injury bracing with rigid cervical collar
Procedure: posterior C1-C2 instrumented fusion — Treatment arm #2 (posterior C1-2 instrumented fusion): Participants randomized to this treatment arm will undergo posterior C1-2 instrumented fusion with either local bone grafting or autologous iliac crest bone grafting with or without allograft bone grafting. Bone grafting decision will be made by the treating surgeon. All remaining decisions surrounding medical and surgical care will be made by the attending spine surgeon involved in each case.
  Arms: posterior C1-2 instrumented fusion

SUMMARY:
This prospective study addresses one of the most controversial topics in the treatment of cervical spine trauma: the management of type II odontoid process fractures in the elderly. It is the hypothesis that surgical treatment will result in improved functional outcome measures, neck pain and mortality rates as compared with nonsurgical management. Furthermore, it is hypothesized that surgical treatment of odontoid process fractures will limit hospital re-admissions and development of medical complications secondary to prolonged immobilization in a cervical orthosis and delayed surgery related to late fracture displacement, which are often associated with non-operative care. Additionally, data from this study will be useful in identifying patient-specific predictors of improved outcome which can be used to optimize treatment algorithms and more effectively counsel patients who sustain these injuries.

ELIGIBILITY:
Inclusion Criteria:

Patients to be considered for trial enrollment will include those:

1. ages 65 and older;
2. presenting with type II odontoid fracture confirmed by CT scan to one of the study centers;
3. deemed appropriate by the attending surgeon involved for C1-2 posterior cervical fusion procedure if surgical management were to be indicated
4. able to independently cooperate in the completion of all study consents, forms and documents.
5. able to speak, read and write English at an elementary school level

Exclusion Criteria:

Patients to be excluded from trial enrolment include:

1. those with previously documented type II odontoid fracture;
2. those with odontoid fracture related to malignancy or infection;
3. those with associated spinal cord injury
4. those with other cervical, thoracic or lumbar injuries requiring surgical intervention
5. those with aberrant/anomalous local anatomy which precludes posterior placement of C1/2 instrumentation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-06-14 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
neck disability | 6 months post randomization
  Measured by validated outcome measure NDI (Neck Disability Index)

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No